CLINICAL TRIAL: NCT06693336
Title: Phase IIa Trial Evaluating the Safety and Therapeutic Effect of SMS001 as an Adjuvant Therapy to Control Tumor Recurrence in Stage Ib-IIIa (N2) Non-Small Cell Lung Cancer (NSCLC) Patients
Brief Title: An Adjuvant Study to Evaluate SMS001 (Paclitaxel) in Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ToLymph Inc. (Industry)
Collaborators: Ozmosis Research Inc. (Industry); University Health Network (UHN) (Unknown); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 132551-1
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung Cancer (NSCLC)
Keywords: NSCLC; Carcinoma
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Confirmation (Experimental): All participants will receive a one-time administration of SMS001 undergoing their scheduled lung cancer surgery. Participants are given SMS001 and are watched very closely for side effects. If the side effects are manageable, then more participants are asked to join the study and are given a higher dose of SMS001, until a pre-defined suitable dose is reached.
  Interventions: Drug: SMS001

INTERVENTIONS:
Drug: SMS001 — One time administration
  Other Names: Paclitaxel

SUMMARY:
This study evaluates the use of SMS001 in patients with lung cancer. SMS001 is a new form of drug Paclitaxel. Doctors want to decide an appropriate safe dose for SMS001 administration, and to see how well it works in treating lung cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To evaluate the safety and tolerability of SMS001 in Non-Small Cell Lung Cancer (NSCLC) patients undergoing cancer surgery.

SECONDARY OBJECTIVES:

1. To evaluate tumor recurrence at 12-month follow-up in NSCLC lung cancer patients treated at a predefined dose.
2. To evaluate disease free survival (DFS) for patients treated with SMS001 at the end of study.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathological confirmed NSCLC
2. Stage Ib, IIa, IIb or IIIa (N2) for both dose escalation and dose confirmation (NOTE: Staging will be according to the AJCC 8th edition)
3. Age ≥18 years and suitable for lung cancer surgery
4. No prior chemotherapy and/or thoracic radiation therapy
5. Normal liver, and renal function at study entry
6. Laboratory requirements:

   1. WBC > 2500/mm3
   2. Neutrophil >1500/mm3
   3. Hemoglobin >10 g/dL
   4. Platelet >100,000/ mm3
   5. AST and ALT < 2.5 x ULN
   6. Total bilirubin < 1.5 x ULN
   7. Creatinine < 2 mg/dL (equivalent to 176.8 μmol/L)
   8. Normal PT/INR and PTT
   9. eGFR >60mL/min/1.73m²
7. QT interval corrected for heart rate using Frederica's formula (QTcF): males < 450msec and females < 470msec
8. Operating surgeon deems patient is candidate for complete surgical resection of lung cancer and lymphadenectomy or lymph node sampling (Wedge resection, segmentectomy or lobectomy are acceptable)
9. Stated willingness to comply with all study procedures and availability for the duration of the study
10. Ability to understand and sign informed consent
11. Women of childbearing potential (WOCBP) must use highly effective methods of contraception for at least 6 months after wafer insertion. Otherwise, women must be postmenopausal (at least 1 y absence of vaginal bleeding or spotting and confirmed by follicle stimulating hormone [FSH] ≥40 mIU/mL [or ≥ 40 IU/L] if less than 2 y postmenopausal) or be surgically sterile. Men must use highly effective methods of contraception for at least 3 months after wafer insertion. Examples of highly effective contraception include: parenteral contraceptives, oral contraceptives, patch contraceptives, implantable hormonal contraceptives, intrauterine device or system, surgical sterilization (hysterectomy, bilateral oophorectomy, and/or bilateral salpingectomy), tubal ligation/occlusion, vasectomized partner, or sexual abstinence, if this is the subject's current practice. Periodic abstinence, i.e., calendar, symptothermal, or post-ovulation methods are not an acceptable form of contraception for this study.

Exclusion Criteria:

If a subject meets any of the following criteria, he/she must be excluded from the study.

1. Evidence of locally advanced T3 or T4 NSCLC or distant metastatic disease.
2. Patients requiring pneumonectomy or sleeve resection.
3. Known sensitivity to any of the study agent components.
4. Patients with a previous malignancy within the last 5 years except non-melanoma skin cancer.
5. Patients receiving induction (neo-adjuvant) chemotherapy and/or radiation prior to surgery.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection. dysfunction of major organ (e.g., liver, kidney etc.), symptomatic congestive heart failure. unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Pregnant or nursing female subjects.
8. Unwilling or unable to follow protocol requirements.
9. Any other condition (e.g., psychiatric disorder) that, in the opinion of the Investigator, may interfere with the patient's ability to comply with the study requirements or visit schedule.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the incidence of treatment-emergent adverse events (Safety and Tolerability) | Day 1 to 52 weeks
  Treatment Emergent Adverse Events included laboratory assessments, physical examination findings, and vital signs.

SECONDARY OUTCOMES:
Incidence of local tumour recurrence | 1 year
  Time from SMS001 treatment to any clinically, histologically or radiologically confirmed local recurrence of NSCLC to mediastinal lymph nodes

OTHER OUTCOMES:
Disease free survival (DFS) | 1 year
  Time from SMS001 treatment to any confirmed recurrence of NSCLC at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhiro Yasufuku MD, PhD, FRCSC, Principal Investigator — University Health Network (UHN)
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No